CLINICAL TRIAL: NCT02654197
Title: Potential Adverse Developmental and Nutritional Consequences of Helicobacter Pylori Infection in Israeli Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-0093-15
Record Dates: First submitted 2015-12-14; First posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-12

CONDITIONS: Helicobacter Pylori Infection; Iron Deficiency Anemia; Child Development
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken for analysis and will be retained for later investigation.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- H.pylori positive children: Healthy children, 6-12 years old, will undergo screening for H. pylori infection by measuring anti-H. pylori and CagA IgG antibodies in the serum. The status of H. pylori infection will be confirmed using breath test (UBT). Children will be classified as i) H. pylori negative, if they test negative on UBT ii) H. pylori positive- CagA negative, if they test positive on UBT, but lack serum CagA IgG antibodies iii) H. pylori positive- CagA positive, if they are positive for H. pylori on UBT and CagA IgG antibodies.
- H.Pylori negative children: Healthy children, 6-12 years old, will undergo screening for H. pylori infection by measuring anti-H. pylori and CagA IgG antibodies in the serum. The status of H. pylori infection will be confirmed using breath test (UBT). Children will be classified as i) H. pylori negative, if they test negative on UBT ii) H. pylori positive- CagA negative, if they test positive on UBT, but lack serum CagA IgG antibodies iii) H. pylori positive- CagA positive, if they are positive for H. pylori on UBT and CagA IgG antibodies.

SUMMARY:
The investigators believe that there is an association between H. pylori infection and nutritional status and between H. pylori infection and cognitive development. The current study will examine this association in Israeli children, aged 6-12 years.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent by parents/guardians and children

Exclusion Criteria:

* Growth retardation history
* History of prior therapy for H. pylori irradiation
* Hematological disorders
* Developmental delays

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children aged 6-12 years residing in the catchment areas of primary care clinics in the Hadera sub-district of Israel.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Changes in means of differences in height | Two years
  The means of the differences in height for age Z score between baseline and follow-up visits
Changes in means of differences in weight | Two years
  The means of the differences in weight for age Z score between baseline and follow-up visits
Changes in means of differences in body mass index | Two years
  The means of the differences in body mass index for age Z score between baseline and follow-up visits

SECONDARY OUTCOMES:
Changes in Iron Biomarkers | Two years
  The means of the differences in iron biomarkers (hemoglobin, ferritin, iron) between baseline and follow-up visits

OTHER OUTCOMES:
Changes in Intelligence quotient (IQ) scores | Two years
  Changes in full-Scale IQ scores and-sub-scores on WISC test between baseline and 24-months follow-up visit: will be defined as the means of the differences of these scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No